CLINICAL TRIAL: NCT04356144
Title: Coagulation Assays in the Critically Ill Patient: a New Approach Using the Thrombomodulin-modified Thrombin Generation Assay (TGA-TM)
Brief Title: Thrombomodulin-modified Thrombin Generation Assay (TGA-TM) in Patients With Critical Infections
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical Scientific Fund of the Mayor of Vienna (Other)
Responsible Party: Principal Investigator, Lukas Infanger, Principal Investigator, Medical University of Vienna
Other Study IDs: TGA-TM-Critical-2019
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Disseminated Intravascular Coagulation; Critical Illness; Sars-CoV2; Viral Infection; Coagulation Disorder, Blood; Covid19
Keywords: TGA; thrombin generation; Sars-CoV2; ROTEM; rotational thromboelastometry; viscoelastic assay; thrombomodulin
MeSH Terms: conditions — Disseminated Intravascular Coagulation; Critical Illness; Virus Diseases; Blood Coagulation Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical infection: Patients with signs of infection with SARS-CoV-2 or already diagnosed infection with SARS-CoV-2 admitted to the ICU
  Interventions: Diagnostic Test: Thrombin Generation Assay (TGA); Diagnostic Test: Thrombomodulin Modified Thrombin Generation Assay (TGA-TM)

INTERVENTIONS:
Diagnostic Test: Thrombin Generation Assay (TGA) — TGA via a fluorimetric module. Coagulation cascade is activated upon addition of different concentrations of tissue factor and phospholipids. The fluorogenic substrate Z-Gly-Gly-Arg-AMC (ZGGR-AMC) is cleaved by formed thrombin over time. By plotting the changes in fluorescence as a function of time (cnt/min), it depicts the "Thrombin Generation Curve" (thrombin generated - plotted against time). The area under the thrombin curve is defined as the endogenous thrombin potential (ETP).
Diagnostic Test: Thrombomodulin Modified Thrombin Generation Assay (TGA-TM) — Recombinant Human Thrombomodulin (TM) is added to the conventional TGA. When recombinant TM is added, the protein C system is fully activated and therefore the ETP obtained reflects both the anti- and procoagulant factors.

SUMMARY:
Inflammation and abnormalities in laboratory coagulation tests are inseparably tied. For example, coagulation abnormalities are nearly universal in septic patients. Coagulation disorders have also been reported in many patients with severe courses of Coronavirus disease 2019 (Covid-19). But it is difficult to assess these changes. Global coagulation tests have been shown to incorrectly assess in vivo coagulation in patients admitted to intensive care units. But other tests are available. Thrombin generation assay (TGA) is a laboratory test which allows the assessment of an individual's potential to generate thrombin. But also in conventional TGA the protein C system is hardly activated because of the absence of endothelial cells (containing natural thrombomodulin) in the plasma sample. Therefore the investigators add recombinant human thrombomodulin to a conventional TGA. Thereby the investigators hope to be able to depict in vivo coagulation more closely than global coagulation tests do.

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU
* Clinical signs of infection with SARS-CoV-2 or already diagnosed infection with SARS-CoV-2
* Neutrophil-Lymphocyte Ratio (NLR) >3

Exclusion Criteria:

* Intake of oral anticoagulants or any kind of parenteral therapeutic anticoagulation prior to ICU admission
* Congenital coagulation disorder
* Treatment with Prothrombin complex concentrate (F. II, VII, IX, X) or activated Prothrombin complex within past 48 hours
* Treatment with recombinant factor VIIa (e.g. eptacog alfa) within past 48 hours
* Treatment with recombinant protein C within past 48 hours
* Active bleeding
* Acute myocardial infarction
* HIV infection
* Chronic pancreatitis
* Liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 critically ill patients with signs of infection with SARS-CoV2 or proven infection with SARS-CoV-2 admitted to Intensive Care Units (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
ETP (AUC) without rhThrombomodulin (rhTM) | 6 months
  nM;
ETP (AUC) with rhThrombomodulin (rhTM) | 6 months
  nM;
ETP-ratio | 6 months
  Ratio of endogenous thrombin potential (ETP) with rhTM to ETP without rhTM
ETP-Normalisation | 6 months
  Comparison of ETP-ratios from ICU patients and ETP-ratios from citrated plasma samples from healthy donors

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided